CLINICAL TRIAL: NCT02591082
Title: A Multi-Center, Post-Marketing, Prospective, Observational Study Following Treatment With Intra-Arterial Delivery of Chemotherapeutic Agents Using the RenovoCath™ RC120 Catheter
Brief Title: Intra-Arterial Treatment of Pancreatic Cancer Using the RenovoCath™ RC120 Catheter
Status: Completed | Type: Observational
Sponsor: RenovoRx (Industry)
Responsible Party: Sponsor
Other Study IDs: RR2
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: RenovoCath™ R120 Catheter — The RenovoCath™ RC120 Catheter will be used to isolate segments of arteries supplying blood to the pancreas. The two balloons on the catheter will be positioned and inflated to temporarily stop blood flow while medication is infused through the catheter between the balloons.

SUMMARY:
This is an observational study to assess patient survival and clinical outcomes after the RenovoCath™ RC120 catheter is used to deliver chemotherapeutic agents to pancreatic tumors.

DETAILED DESCRIPTION:
This is an observational, registry study to assess patient survival and clinical outcomes of the RenovoCath™ RC120 catheter when used to deliver chemotherapeutic agents to pancreatic tumors. Blood samples will be drawn in a subset of patients to assess the systemic concentration of the chemotherapeutic agent.

The RenovoCath™ RC120 Catheter is an endovascular multi-lumen, two-handled catheter designed to isolate variable segments of arteries supplying the target organ using two slideable, compliant balloons. Upon inflation of the proximal occlusion balloon and the distal occlusion balloon, the catheter may isolate the selected site to specifically deliver radiopaque and therapeutic agents including, but not limited to chemotherapeutic drugs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Diagnosed with unresectable or borderline resectable pancreatic adenocarcinoma confirmed by histology or cytology
* Without current myelotoxicity and with sufficient health status to undergo a catheterization procedure
* Willing to provide informed consent and comply with the required follow-up.

Exclusion Criteria:

* Have received prior chemotherapy and/or radiation therapy within 14 days prior to the first intra-arterial treatment.
* Currently participating in another active drug or device study or registry protocol that would interfere with this study.
* Vulnerable populations: prisoners, pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with unresectable or borderline resectable pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-12; Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Survival | 2 Years
  Duration of survival in patients diagnosed with pancreatic cancer who undergo intra-arterial delivery of chemotherapeutic agents to the pancreas

SECONDARY OUTCOMES:
Tumor response | 6 months
  Time to tumor response in the primary site of application as assessed by imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Ramtin Agah, MD, Study Director — Chief Medical Officer
Locations (5):
- United States (5):
  - Good Samaritan Hospital, San Jose, California
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - Florida Hospital, Tampa, Florida
  - Montefiore Hospital, The Bronx, New York
  - East Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hatoum H, Rosemurgy A 2nd, Bastidas JA, Zervos E, Muscarella P 2nd, Edil BH, Cynamon J, Johnson DT, Thomas C, Swinson BM, Nordgren A, Vitulli P, Nutting C, Gipson M, Tsobanoudis A, Agah R. Treatment of locally advanced pancreatic cancer using localized trans-arterial micro perfusion of gemcitabine: combined analysis of RR1 and RR2. Oncologist. 2024 Aug 5;29(8):690-698. doi: 10.1093/oncolo/oyae178. PMID 39049803